CLINICAL TRIAL: NCT05147688
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Pulmonary Diseases
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for Pulmonary Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-1-MSC-013
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Disease; Asthma; Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Disease; Asthma; stem cell treatment; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Pulmonary Diseases

DETAILED DESCRIPTION:
In this patient funded trial, patients with pulmonary disease will receive a single intravenous infusion of UC-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary disease
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: Forced vital capacity (FVC) | Four year follow-up
  It will be completed for each follow up point.
Efficacy: Pulmonary function test | Four year follow-up
  It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Averyanov A, Koroleva I, Konoplyannikov M, Revkova V, Lesnyak V, Kalsin V, Danilevskaya O, Nikitin A, Sotnikova A, Kotova S, Baklaushev V. First-in-human high-cumulative-dose stem cell therapy in idiopathic pulmonary fibrosis with rapid lung function decline. Stem Cells Transl Med. 2020 Jan;9(1):6-16. doi: 10.1002/sctm.19-0037. Epub 2019 Oct 15. PMID 31613055
- [Background] Fishman JE, Kim GJ, Kyeong NY, Goldin JG, Glassberg MK. Intravenous stem cell dose and changes in quantitative lung fibrosis and DLCO in the AETHER trial: a pilot study. Eur Rev Med Pharmacol Sci. 2019 Sep;23(17):7568-7572. doi: 10.26355/eurrev_201909_18877. PMID 31539148
- [Background] Cruz FF, Borg ZD, Goodwin M, Sokocevic D, Wagner D, McKenna DH, Rocco PR, Weiss DJ. Freshly thawed and continuously cultured human bone marrow-derived mesenchymal stromal cells comparably ameliorate allergic airways inflammation in immunocompetent mice. Stem Cells Transl Med. 2015 Jun;4(6):615-24. doi: 10.5966/sctm.2014-0268. Epub 2015 Apr 29. PMID 25925837
- [Background] Trzil JE, Masseau I, Webb TL, Chang CH, Dodam JR, Liu H, Quimby JM, Dow SW, Reinero CR. Intravenous adipose-derived mesenchymal stem cell therapy for the treatment of feline asthma: a pilot study. J Feline Med Surg. 2016 Dec;18(12):981-990. doi: 10.1177/1098612X15604351. Epub 2015 Sep 17. PMID 26384398